CLINICAL TRIAL: NCT01817907
Title: The Effects of Trazodone on the Severity of Obstructive Sleep Apnea
Brief Title: The Effects of Trazodone on Sleep Apnea Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BWH-2009P001862; P01HL095491-01A1 (NIH)
Record Dates: First submitted 2012-11-22; First posted 2013-03-26 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Apnea- Hypopnea index; Arousal Threshold
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Sugars; Trazodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive a sugar pill during their placebo night sleep study.
  Interventions: Drug: Placebo pill
- Trazodone (Active Comparator): Subjects will receive trazodone during their treatment night sleep study
  Interventions: Drug: Trazodone

INTERVENTIONS:
Drug: Placebo pill — Subjects will receive a sugar pill during the placebo arm
  Other Names: Sugar pill
  Arms: Placebo
Drug: Trazodone — Subjects will receive trazodone during one of their treatment arm studies
  Arms: Trazodone

SUMMARY:
In Obstructive sleep apnea (OSA), the upper airway closes over and over again during sleep. This leads to disrupted sleep (waking up during the night), daytime sleepiness, and an increased risk for developing high blood pressure. Currently, the best treatment for obstructive sleep apnea is sleeping with a mask that continuously blows air into the nose (i.e. Continuous positive airway pressure [CPAP] treatment). While CPAP treatment stops the upper airway from closing in most people, many people have difficulty sleeping with the mask in place and therefore do not use the CPAP treatment. This research study is being conducted to learn whether using a sedative will improve OSA severity by altering some of the traits that are responsible for the disorder.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repetitive collapse or 'obstruction' of the pharyngeal airway during sleep. These obstructions result in repetitive hypopneas/apneas and intermittent hypoxia/hypercapnia, as well as surges in sympathetic activity. Such processes disturb normal sleep and impair neurocognitive function, often resulting in excessive daytime sleepiness and decreased quality of life. Furthermore, OSA is associated with cardiovascular morbidity and mortality, making OSA a major health concern.

Current evidence suggests that OSA pathogenesis involves the interactions of at least four physiological traits comprising: 1) the pharyngeal anatomy and its propensity towards collapse. This collapsibility of the upper airway is measured as the critical closing pressure or PCRIT. 2) the ability of the upper airway dilator muscles to activate and reopen the airway during sleep (i.e. neuromuscular compensation) measured as the increase in upper airway electromyography (EMG) activity above the baseline level. 3) the arousal threshold from sleep (i.e. the propensity for hypopneas/apneas to lead to arousal and fragmented sleep) measured as the epiglottic pressure occurring just at the time of arousal and 4) the stability of the ventilatory feedback loop (i.e. loop gain). Continuous positive airway pressure (CPAP) is the most common treatment for OSA but it is often poorly tolerated; only ~50% of patients diagnosed with OSA continue therapy beyond 3 months. Given this limitation, alternative approaches have been tested and have generally focused on the use of oral appliances and upper airway surgery.

In addition to these alternative therapies, the use of pharmacological agents for the treatment of OSA has been gaining widespread interest. Previous data have shown that the non-myorelaxant hypnotic trazodone increases the arousal threshold however its effects on sleep apnea severity remain unclear. Based on studies showing that increasing the arousal threshold with a different hypnotic improves sleep apnea severity, we hypothesize that trazodone will increase the arousal threshold and this will be associated with an improvement in sleep apnea severity.

Therefore the overall aim of this study is to examine the effects that trazodone has on OSA severity.

STUDY DESIGN:

A double-blinded randomized control design will be used. Initially, participants will be randomized to the trazodone or placebo arm where they will have both a clinical polysomnography (PSG) with the addition of an epiglottic pressure cathether. The purpose of the clinical PSG is to determine the severity of OSA (i.e. AHI) and the epiglottic catheter allows the calculation of the arousal threshold to be completed.

During the trazodone arm, participants will be given trazodone (100mg by mouth) to take before bed. During the placebo arm, subjects will be given a placebo to take before bed.

Participants will have at least a 1-week washout period before cross over to the next arm of the study whereby the clinical PSG will be repeated. In total each subject will be studied for 2 nights.

ELIGIBILITY:
Inclusion Criteria for OSA Patients:

* OSA (elevated AHI).
* Age range 18-70 years.

Exclusion Criteria:

* Any known cardiac (apart from treated hypertension), pulmonary (including asthma), renal, neurologic (including epilepsy), neuromuscular, or hepatic disease.
* Susceptible to stomach ulcers.
* Pregnant women.
* History of hypersensitivity to Afrin, Lidocaine, trazodone and/or donepezil.
* History of bleeding diathesis and/or gastrointestinal bleeding.
* Use of any medications that may affect sleep or breathing.
* A psychiatric disorder, other than mild depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Substantial cigarette (>5/day), alcohol (>3oz/day) or use of illicit drugs.
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day.
* Desaturations to below 70% lasting greater than 10 seconds in duration per event on polysomnography.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Smales ET, Edwards BA, Deyoung PN, McSharry DG, Wellman A, Velasquez A, Owens R, Orr JE, Malhotra A. Trazodone Effects on Obstructive Sleep Apnea and Non-REM Arousal Threshold. Ann Am Thorac Soc. 2015 May;12(5):758-64. doi: 10.1513/AnnalsATS.201408-399OC. PMID 25719754

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First: Subjects will receive a sugar pill (placebo) during their first sleep study night and will receive a pill of trazodone (100 mg) during their second sleep study night.
- Trazodone First: Subjects will receive a pill of trazodone (100 mg) during their first sleep study night and will receive a sugar pill (placebo) during their second sleep study night.
Period: First Intervention
Arm/Group | Placebo First | Trazodone First
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Placebo First | Trazodone First
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First | Trazodone First
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo First: Subjects will receive a sugar pill during their placebo night sleep study.
  Placebo pill: Subjects will receive a sugar pill during the placebo arm
- Trazodone First: Subjects will receive trazodone during their treatment night sleep study
  Trazodone: Subjects will receive trazodone during one of their treatment arm studies
- Total: Total of all reporting groups
Arm/Group | Placebo First | Trazodone First | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (7) | 53 (14) | 53 (10)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index
Description: The Apnea-Hypopnea Index (AHI) is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow).
Time Frame: Participants will be assessed on 2 nights over an average period of 2 weeks.
Population: two subjects were excluded from analysis because of excessive number of artifacts
Measure: Mean (Standard Error); unit: events/hour
Arm/Group | Placebo | Trazodone
Number analyzed (Participants) | 13 | 13
events/hour | 38.7 (6.2) | 28.5 (5.6)

2. Secondary Outcome: Arousal Threshold (cmH2O)
Description: Subjects will have an epiglottic pressure catheter placed during their sleep studies. We will use the swing in the epiglottic pressure trace just prior to arousal to calculate the respiratory drive stimulus that is associated with an a respiratory induced arousal.
Time Frame: Participants will be assessed on 2 nights over an average period of 2 weeks.
Population: two subjects were excluded from analysis because of excessive number of artifacts
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Placebo | Trazodone
Number analyzed (Participants) | 13 | 13
cmH2O | -19.3 (3.9) | -20.3 (3.7)
Statistical Analysis 1: Comparison: Placebo vs Trazodone; Test type: Superiority or Other; p = 0.52, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo | Trazodone
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No